CLINICAL TRIAL: NCT03420430
Title: Use of GL-ONC1 in Patients With Advanced Cancers With No Standard of Care
Brief Title: Expanded Access to Provide GL-ONC1 for the Treatment of Advanced Cancers With No Standard of Care
Status: No longer available | Type: Expanded Access
Sponsor: Genelux Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: GL-ONC1-021
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Advanced Stage Cancer (Solid Tumor Disease for 4 Patients); Acute Myeloid Leukemia (6 Patients)
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: GL-ONC1

SUMMARY:
GL-ONC1 expanded access is for patients who are ineligible for an ongoing GL-ONC1 clinical trial. Expanded access is intended to treat individual patients with advanced stage cancers, including blood cancer, with no standard of care options for treatment. Potential patients will be evaluated individually depending on GL-ONC1 product supply.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced cancers with no standard of care option for treatment.
* Willing and able to provide written, signed informed consent.
* Use of adequate contraception.
* Negative pregnancy test.

Exclusion Criteria:

* Have not recovered from severe adverse events from prior therapy.
* Major surgery occurred within 28 days prior to treatment.
* Known immune system disorders such as HIV, or active hepatitis B or C infection.
* Clinically significant cardiac disease (New York Heart Association Class III or IV).
* Have received prior therapy with an oncolytic virus of any type.
* Be receiving antiviral agent active against vaccinia virus (e.g., cidofovir, vaccinia immunoglobulin, imatinib, ST-246).
* Have known allergy to ovalbumin or other egg products.
* Have clinically significant dermatological disorders (e.g., eczema, psoriasis, or any unhealed skin wounds or ulcers) as assessed by the treating physician.

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Florida Hospital Cancer Institute, Orlando, Florida, United States

REFERENCES:
- See also: Sponsor website — http://www.genelux.com